CLINICAL TRIAL: NCT01126268
Title: Twice Daily Altabax Application for the Treatment of Uncomplicated Soft Tissue Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Adelaide Hebert, Professor of Dermatology and Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-09-0650
Record Dates: First submitted 2010-04-19; First posted 2010-05-19 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Impetigo; Folliculitis; Secondarily Infected Eczema; Minor Soft Tissue Infections
Keywords: Eczema; Atopic dermatitis; Infection; Impetigo; Folliculitis
MeSH Terms: conditions — Impetigo; Folliculitis; Eczema; Dermatitis, Atopic; Infections | interventions — retapamulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retapamulin ointment 1% (Experimental)
  Interventions: Drug: Retapamulin (Altabax)

INTERVENTIONS:
Drug: Retapamulin (Altabax) — Retapamulin ointment, applied topically twice daily for five days
  Other Names: Altabax

SUMMARY:
The purpose of this study is to document the clinical and bacteriological efficacy of retapamulin in the treatment of subjects with bacterial infections, including impetigo, folliculitis, and minor soft tissue infections including secondarily infected eczema presumed to be caused by methicillin resistant Staph aureus. Male and female patients ages 9 months to 98 years will be recruited from a university based dermatology clinic. Upon enrollment, wound cultures will be collected, and then subjects will apply topical retapamulin twice daily for five days. The primary endpoint will be resolution of methicillin-resistant Staphylococcus aureus (MRSA) infection based on clinical presentation and physical exam, as well as bacteriological efficacy based on culture results. It is anticipated that approximately 75 patients will be enrolled, with expectation that approximately 50 of these patients will have MRSA infections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients from 9 months of age up to 98 years of age.
* Clinical diagnosis of impetigo, folliculitis, or minor soft tissue infection including secondarily infected eczema presumed to be caused by Staphylococcus aureus.
* The patient, and if applicable the parent or guardian, is able to give informed consent
* Females of child bearing potential have a negative urine pregnancy test.
* Patient, and if applicable parent or guardian, are willing to and capable of complying with the study protocol.

Exclusion Criteria:

* Subject who has used a topical antibacterial medication to the area being treated within the last 48 hours.
* Subject who has been enrolled in a clinical trial within the last 30 days.
* Subject with signs of systemic infection (such as fever), or with evidence of abscess or cellulitis at the site to be treated.
* Subject has a bacterial skin infection which would not be appropriately treated by a topical antibiotic in the opinion of the investigator
* Subjects who have taken oral antibiotics within the last 7 days.
* Subjects with known sensitivity to the study medication.
* The subject is pregnant or breastfeeding

Ages: 9 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide A Hebert, M.D., Principal Investigator — University of Texas Health Science Center at Houston Department of Dermatology
Locations (1):
- Houston Medical Center Building, Houston, Texas, United States

REFERENCES:
- [Result] Bohaty BR, Choi S, Cai C, Hebert AA. Clinical and bacteriological efficacy of twice daily topical retapamulin ointment 1% in the management of impetigo and other uncomplicated superficial skin infections. Int J Womens Dermatol. 2015 Mar 2;1(1):13-20. doi: 10.1016/j.ijwd.2014.12.002. eCollection 2015 Feb. PMID 28491950

RESULTS

PARTICIPANT FLOW:
Groups:
- Retapamulin Ointment 1% Group: Subjects with clinically diagnosed with impetigo, folliculitis, or minor soft tissue infection suitable for treatment with a topical antibiotic were screened, and if qualified, they received topical retapamulin ointment 1% twice daily for 5 days.
Period: Overall Study
Arm/Group | Retapamulin Ointment 1% Group
Started | 38
Completed | 37
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (25.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Wound Cultures Were Positive for MRSA and Who Were Determined to be a Clinical Success at the Follow-up Visit
Description: Clinical success is defined as no further signs or symptoms of infection present, including erythema, purulence, crusting, edema, warmth and pain.
Time Frame: 6 to 8 days after treatment
Population: Participants whose wound cultures were positive for MRSA
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 7
participants | 5

2. Secondary Outcome: Clinical Response at Follow up as Assessed by a Rating Scale
Description: Clinical response was based on clinical evaluation by the investigator at the follow-up visit using a predefined scale with the following categories: (1) clinical success, (2) clinical improvement, (3) no change, (4) clinical failure, and (5) unable to determine. Patients who were designated as clinical success as defined in number 1 above were considered a true "clinical success" while all others were considered a "clinical failure." Patients were classified with an outcome of "unable to determine" if they missed their follow-up visit or refused clinical examination.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  1. Clinical success | 23
  2. Clinical improvement | 11
  3. No change | 0
  4. Clinical failure | 1
  5. Unable to determine | 0

3. Secondary Outcome: Microbiologic Response at Follow up as Assessed by a Rating Scale
Description: Microbiological response was determined by the investigator at the follow-up visit using the following microbiological outcomes: (1) microbological eradication, (2) presumed microbiological eradication, (3) presumed microbiological improvement, (4) microbiological persistence, (5) presumed microbiological persistence, (6) unable to determine, (7) new pathogen, and (8) colonization. Patients who were designated microbiological eradication, presumed microbiological eradication, presumed microbiological improvement, or colonization as defined in numbers 1, 2, 3, and 8 above were considered a "microbiological success" while all others were considered "microbiological failure."
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  1. Microbiological eradication | 1
  2. Presumed microbiological eradication | 23
  3. Presumed microbiological improvement | 10
  4. Microbiological persistence | 1
  5. Presumed microbiological persistence | 0
  6. Unable to determine | 0
  7. New pathogen | 0
  8. Colonization | 0

4. Secondary Outcome: Number of Participants Who Were a Therapeutic Success
Description: Therapeutic response was determined from the clinical response and the microbiological response. Patients who qualified as both a "clinical success" and a "microbiological success" were deemed a "therapeutic success," and all others were deemed "therapeutic failures."
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants | 23

5. Secondary Outcome: Erythema (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 0
  Minimal | 10
  Moderate | 25
  Severe | 0

6. Secondary Outcome: Erythema (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 9
  Minimal | 24
  Moderate | 2
  Severe | 0

7. Secondary Outcome: Purulence (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 10
  Minimal | 14
  Moderate | 10
  Severe | 1

8. Secondary Outcome: Purulence (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 34
  Minimal | 1
  Moderate | 0
  Severe | 0

9. Secondary Outcome: Crusting (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 2
  Minimal | 8
  Moderate | 23
  Severe | 2

10. Secondary Outcome: Crusting (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 25
  Minimal | 9
  Moderate | 1
  Severe | 0

11. Secondary Outcome: Tissue Edema (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 3
  Minimal | 19
  Moderate | 13
  Severe | 0

12. Secondary Outcome: Tissue Edema (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 19
  Minimal | 16
  Moderate | 0
  Severe | 0

13. Secondary Outcome: Tissue Warmth (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 9
  Minimal | 20
  Moderate | 6
  Severe | 0

14. Secondary Outcome: Tissue Warmth (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 21
  Minimal | 14
  Moderate | 0
  Severe | 0

15. Secondary Outcome: Pain (Sign and Symptom of Infection) at Baseline
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 8
  Minimal | 19
  Moderate | 8
  Severe | 0

16. Secondary Outcome: Pain (Sign and Symptom of Infection) at Follow up
Description: Signs and symptoms of infection were classified as one of the following: absent, minimal, moderate, or severe.
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
participants
  Absent | 26
  Minimal | 9
  Moderate | 0
  Severe | 0

17. Secondary Outcome: Wound Size at Baseline
Description: Wound size area was determined by measuring the greatest length of the wound in two perpendicular dimensions with a standard metric ruler. The two measurements were multiplied together to provide an estimate of the overall wound size. Surrounding erythema was not included in the measurement.
Time Frame: baseline
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
cm^2 | 14.43 (25.38)

18. Secondary Outcome: Wound Size at Follow up
Description: as for outcome 17
Time Frame: 6 to 8 days after treatment
Population: All participants who had a pathogen isolated from the treatment area at baseline upon microbiological testing
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 35
cm^2 | 4.31 (17.71)

19. Secondary Outcome: Number of Participants Reporting Any Adverse Event (AE)
Description: AEs included burning at application site, upper respiratory infection, furuncle, cough, and a rash at a site other than the application site. See the Adverse Events section for more detailed information.
Time Frame: baseline to 6 to 8 days after treatment
Population: All participants who received at least 1 dose of Retapamulin (Altabax)
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment 1%
Number analyzed (Participants) | 38
participants | 4

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Retapamulin Ointment 1%
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retapamulin Ointment 1% (N=38)
Burning at Retapamulin (Altabax) application site (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Rash at site other than the Retapamulin (Altabax) application site (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No